CLINICAL TRIAL: NCT07336498
Title: Clinical Evaluation and Cone Beam Computed Tomography Analysis of Amniotic Membrane, Putty Mineral Trioxide Aggregate and Biodentine as Therapeutic Agents for Apexogenesis of Immature Permanent Molars: A Randomized Clinical Trial
Brief Title: Clinical Evaluation and Cone Beam Computed Tomography Analysis of Different Biomaterials for Apexogenesis of Immature Permanent Molars
Acronym: MTA/CBCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Ezz Eldeen Ghareep, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 1163/6935
Record Dates: First submitted 2025-11-29; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Vital Pulp Therapy in Young Permanent Tooth

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Biodentine will be placed directly in the pulp chamber (Experimental)
  Interventions: Procedure: Vital pulp therapy of immature permanent teeth
- Previously trimmed amniotic membrane will be placed directly in the pulp chamber (Experimental)
  Interventions: Procedure: Vital pulp therapy of immature permanent teeth
- Putty MTA will be placed directly in the pulp chamber (Other)
  Interventions: Procedure: Vital pulp therapy of immature permanent teeth

INTERVENTIONS:
Procedure: Vital pulp therapy of immature permanent teeth — Conventional access cavity will be done with a high-speed bur using copious water spray. The coronal pulp amputation will be performed using a sharp spoon excavator. In order to achieve hemostasis sterilized cotton pellet moistened with sterile saline will be placed over the pulp's stumps for 5 minutes, followed by application of the therapeutic agent. The prepared cavities of all molars will be sealed with a layer of glass ionomer over the therapeutic agents and subsequently will be covered with composite resin restoration.

SUMMARY:
The present study will be conducted to clinically evaluation and cone beam computed tomography analysis of amniotic membrane, putty mineral trioxide aggregate and biodentine as therapeutic agents for apexogenesis of immature permanent molars

DETAILED DESCRIPTION:
An immature permanent tooth is defined as, a newly erupted permanent tooth with incomplete root apex formation. Since root development is completed in 2-3 years after tooth eruption into the oral cavity, loss of pulp vitality in the immature permanent tooth affected by caries, traumatic injury, or other causes creates major problems. The primary goal of pulp therapy is to maintain the integrity of the teeth while maintaining the vitality of the pulp, especially in young permanent teeth with immature roots to enhance root dentin formation. An increasingly popular therapy option for pulp damage in immature permanent molars is apexogenesis. Vital pulp therapy involves the complete removal of the coronal pulp and the placement of an acceptable material into the pulp chamber. With the invention of calcium silicate material namely mineral trioxide aggregate (MTA), it became preferred to calcium hydroxide in the treatment of exposed pulp. MTA demonstrated excellent biocompatibility, low solubility, outstanding sealing properties and antibacterial effect. However, MTA has some limitations regarding the long setting time and difficult handling. Premixed calcium silicate cements were developed to facilitate manipulation with no need for mixing, such as using the putty formulation which allows better handling with a thicker consistency Additionally, Biodentine was introduced as a tricalcium silicate-based bioceramic, with comparable physical properties to dentine, thus, it is also called dentine replacement material and has applications like those of MTA. Considering the limitations of MTA, biodentine has been developed with enhanced physicochemical properties such as a fast-setting time with an initial setting time between 9 and 12 minutes due to the presence of calcium chloride. Its short setting time allows restoration to be made in one session with easier chairside handling than MTA. Recently, novel biologically based material has been developed from the innermost layer of the placenta with highly rich stem cell reservoirs and is called amniotic membrane. The amniotic membrane is rich in growth factors, various types of collagens (such as types I, III, IV, V, and VII), along with proteoglycans, elastin and hyaluronic acid. It possesses a range of beneficial properties, including anti-inflammatory, antimicrobial and analgesic which make it a unique option for wound healing, providing a supportive environment that promotes the survival and proliferation of mesenchymal progenitor cells. In dentistry, researchers supported its application in regenerative endodontic therapy by providing a growth factors that promote stem cell growth and formation of a new dentine-pulp complex. Therefore, in the present study, clinical and radiographic evaluation will be done to assess the effectiveness of different biomaterials in managing immature permanent tooth with pulp exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients without any systemic disease aged 7 to 10 years old.
* Vital immature permanent molars with deep carious lesions.
* Restorable tooth
* No clinical signs and symptoms of irreversible pulpitis including spontaneous pain, tenderness to percussion, swelling or sinus tract.
* No radiographic evidence of periapical abscess, internal or external resorption.

Exclusion Criteria:

* Patients with known allergies to any of the dental materials to be used.
* Bleeding could not be controlled within 5 minutes after complete pulpotomy
* Teeth with root fractures
* Carious furcation involvement

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes | Base line, 7 days, 3 months, 6 months , 12 months
  Clinical assessment of the treated immature molars in each follow up period as follow:
  1. Presence or Absence of pain or sensitivity to percussion.
  2. Presence or absence of any evidence of swelling, or sinus tract.
  3. Presence or absence of excessive mobility of the treated teeth .

SECONDARY OUTCOMES:
Radiographic assessment of root length by CBCT | Baseline (immediately post-operative ) and 12 months post-operative
  The CBCT scanning was performed immediately after treatment to serve as the baseline and at 12 months follow-up periods to evaluate changes in the root for each tooth in all groups.
  Root length: the sagittal section was used to measure the root length for each root using the CBCT ruler to draw a line from the center point of the line connecting CEJ to the most apical point in the center of the root apex.
  the percentage of increase in root length of the immature permanent molar was calculated by the following formula: (12 months value-baseline value)/(Preoperative value) ×100
Radiographic assessment of diameter of apical foramen by CBCT | Baseline (immediately post-operative) and 12 months post-operative)
  At the most apical point buccolingually in the sagittal view of the CBCT, the diameter of the apical foramen was measured using the CBCT ruler for each root of the immature permanent tooth. The percentage reduction of the apical diameter was calculated using this formula:
  (baseline value-12 months value)/(Preoperative value)×100
Radiographic assessment of radiographic root area by CBCT | Baseline(immediately post-operative) and at 12 months post-operative
  Using the CBCT polygon selection tool at the sagittal section and below a straight line marking the cementoenamel junction, the root area was outlined from the surrounding periodontal environment. The pulp space area was then calculated using the same technique, tracing the reference points around the pulp space with the polygon tool. Finally, the pulp space area was subtracted from the outer root area to determine the radiographic root area. The percentage of increase in radiographic root area of the immature permanent molar was calculated by the following formula:
  (12 months value-baseline value)/(Preoperative value) ×100

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al-Azhar University, Cairo (Boys Branch), Cairo, Egypt

REFERENCES:
- [Background] Duncan HF, Nagendrababu V, El-Karim IA, Dummer PMH. Outcome measures to assess the effectiveness of endodontic treatment for pulpitis and apical periodontitis for use in the development of European Society of Endodontology (ESE) S3 level clinical practice guidelines: a protocol. Int Endod J. 2021 May;54(5):646-654. doi: 10.1111/iej.13501. Epub 2021 Mar 15. PMID 33630330
- [Background] Dentistry AAoP. Pulp therapy for primary and immature permanent teeth. The Reference Manual of Pediatric Dentistry Chicago, Ill: American Academy of Pediatric Dentistry. 2021;399407.